CLINICAL TRIAL: NCT04304183
Title: Defecation Function and Quality of Life in the Patients Treated With Surgery for Slow Transit Constipation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Third Military Medical University (Other)
Responsible Party: Principal Investigator, Weidong Tong, Professor, Third Military Medical University
Other Study IDs: 20190410
Record Dates: First submitted 2019-05-06; First posted 2020-03-11 (Actual); Last update posted 2023-11-27 (Actual); Status verified 2023-11

CONDITIONS: Defecation Function; Quality of Life
Keywords: Slow transit constipation; Defecation function; Quality of life

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- slow transit constipation: patients diagnosed with slow transit constipation had undergone surgery.
  Interventions: Procedure: total colectomy, ileorectal anastomosis

INTERVENTIONS:
Procedure: total colectomy, ileorectal anastomosis — all patients underwent total colectomy and ileorectal anastomosis.The anastomosis was stapled in all patients.

SUMMARY:
Although surgical options for slow transit constipation (STC) have been proven to be a definite treatment, improvements in the associated defecation function and quality of life are rarely studied. This study aims to investigate the effectiveness of total or subtotal colectomy, with respect to short- and long-term defecation function and overall quality of life in 5-year regular follow-up.

DETAILED DESCRIPTION:
Constipation is an ever-growing problem and one of the most common gastrointestinal symptoms, affecting 10-15% of adults in the USA and 8.2% of the general population in China. Slow-transit constipation, representing 15~30% constipated patients, is characterized by a loss in the colonic motor activity. Factors such as increasing age, female sex, physical inactivity, endocrine, metabolism, neurological factors, drug use, and depression are associated with constipation. While most patients with constipation are mild and treated easily by a behavioral and medical way, a minority of patients suffering from long-term intractable symptoms and poor quality of life and showing no response to any medical interventions are ultimately recommended for surgery.

Since the effectiveness of colectomy for constipation was first reported by Lane a century ago, surgical treatment for constipation has been greatly developed[6], including ileorectal anastomosis (IRA), cecorectal anastomosis(CRA), colonic exclusion, antegrade enemas (the Malone procedure), modified Duhamel surgery, and permanent ileostomy. Currently, the main surgical procedures for STC are IRA and CRA, which have been widely confirmed to increase bowel-movement frequency in a huge number of patients. However, the reported outcomes of colectomy are controversial and conflicting.In these studies, lack of prospectively defined follow-up intervals is a general problem. Moreover, long-term outcomes of surgery for STC are rarely reported. Furthermore, negatively persistent symptoms including abdominal pain, bloating, intractable diarrhea, malnutrition, constipation recurrence, fecal incontinence, and intestinal obstruction are not uncommon following surgery, adversely affecting defecation function and quality of life following these procedures.

This study aims to investigate the effectiveness of total or subtotal colectomy, with respect to short- and long-term defecation function and overall quality of life during 5-year regular follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. The clinical manifestations all met the Roman IV standard for the diagnosis of functional constipation.
2. Patients with severe constipation symptoms were unable to defecate naturally and need laxatives to assist defecation or still unable to defecate.
3. Colonic transport tests showed that the opaque X-ray markers remained more than 20% after 72 hours.
4. All conservative treatment for more than 1 year failed.
5. Patients had a strong desire for surgery, and no other contraindications to surgery.

Exclusion Criteria:

1. Megacolon was detected with barium enema examination.
2. Colonoscopy suggested the presence of intestinal organic lesions or a history of colorectal cancer treatment.
3. Gastric and small intestinal transport dysfunction.
4. There are depression, anxiety and other mental symptoms.
5. Constipation type irritable bowel syndrome.
6. History of inflammatory bowel disease.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients diagnosed with STC in the investigator's department were preoperatively included.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
The number of bowel movements | from the pre-operation to the five years following surgery
  the number of bowel movements will be recorded in terms of times per week.
The scales of Wexner Constipation | from the pre-operation to the five years following surgery
  the scales of Wexner Constipation will be recorded in terms of scores.
The scales of Wexner Incontinence | from the pre-operation to the five years following surgery
  the scales of Wexner Incontinence will be recorded in terms of scores.
The incidence of abdominal pain | from the pre-operation to the five years following surgery
  the incidence of abdominal pain will be recorded in terms of percent.
The incidence of bloating | from the pre-operation to the five years following surgery
  the incidence of bloating will be recorded in terms of percent.
The incidence of diarrhea | from the pre-operation to the five years following surgery
  the incidence of diarrhea will be recorded in terms of percent.
The incidence of straining | from the pre-operation to the five years following surgery
  the incidence of straining will be recorded in terms of percent.
The incidence of laxative | from the pre-operation to the five years following surgery
  the incidence of laxative will be recorded in terms of percent.
The incidence of enema use | from the pre-operation to the five years following surgery
  the incidence of enema use will be recorded in terms of percent.
The scales of Gastrointestinal Quality of Life Index | from the pre-operation to the five years following surgery
  the scales of Gastrointestinal Quality of Life Index will be recorded in terms of scores.
The short-form(SF)-36 survey | from the pre-operation to the five years following surgery
  There are eight spheres in the SF-36 survey, including physical function, role physical, role emotional, physical pain, vitality, mental health, social function and general health. Results of each sphere will be recorded in terms of scores.

SECONDARY OUTCOMES:
Number of Participants with complications | from the pre-operation to the five years following surgery
  Postoperative complications includes short-term and long-term complications, such as ileus, anastomotic leak, small intestinal obstruction, constipation recurrence and so on. Number of Participants with complications will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Weidong Tong, MD, Study Chair — Army Military Medical University
Locations (1):
- Weidong Tong, Yuzhong, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Wei D, Cai J, Yang Y, Zhao T, Zhang H, Zhang C, Zhang Y, Zhang J, Cai F. A prospective comparison of short term results and functional recovery after laparoscopic subtotal colectomy and antiperistaltic cecorectal anastomosis with short colonic reservoir vs. long colonic reservoir. BMC Gastroenterol. 2015 Mar 18;15:30. doi: 10.1186/s12876-015-0257-7. PMID 25887580
- [Result] Macha MR. The feasibility of laparoscopic subtotal colectomy with cecorectal anastomosis in community practice for slow transit constipation. Am J Surg. 2019 May;217(5):974-978. doi: 10.1016/j.amjsurg.2019.03.018. Epub 2019 Mar 26. PMID 30948148